CLINICAL TRIAL: NCT00175903
Title: A Therapeutic Confirmatory, Open-label, Multi-center, Randomized 2 Parallel Groups, Community-based Trial Studying the Efficacy and Safety of Levetiracetam (1000 to 3000 mg/Day Oral Tablets 250-500 mg b.i.d.) Compared to Sodium Valproate (1000 to 2000 mg/Day Oral ER Tablets 300-500 mg b.i.d.) and Carbamazepine (600 to 1600 mg/Day Oral CR Tablets 200-400 mg b.i.d.) as Monotherapy in Subjects With Newly Diagnosed Epilepsy.
Brief Title: Levetiracetam Versus Standard Antiepileptic Drugs (Carbamazepine and Valproate) Used as Monotherapy in Patients With Newly Diagnosed Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N01175; 2004-001339-41 (EudraCT Number)
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Epilepsy
Keywords: Newly Diagnosed Epilepsy; Levetiracetam; Keppra; Carbamazepine; Valproate
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (Experimental): Daily dose of 1000 to 3000 mg film-coated oral tablets, 250-500 mg twice daily.
  Interventions: Drug: Levetiracetam
- Older Antepileptic Drugs (Active Comparator): Older AEDs consist of CBZ-CR 200 mg and 400 mg and VPA-ER 300 mg and 500 mg.
  Interventions: Drug: Carbamazepine Controlled Release (CBZ-CR); Drug: Valproate Extended Release

INTERVENTIONS:
Drug: Levetiracetam — Daily dose of 1000 to 3000 mg film-coated oral tablets, 250-500 mg twice daily.
  Arms: Levetiracetam
Drug: Carbamazepine Controlled Release (CBZ-CR) — Daily dose of 600-1600 mg CR oral tablets, 200 mg and 400 mg twice daily.
  Arms: Older Antepileptic Drugs
Drug: Valproate Extended Release — Daily dose of 1000-2000 mg ER oral tablets, 300 mg and 500 mg twice daily.
  Arms: Older Antepileptic Drugs

SUMMARY:
Study N01175 was to compare overall effectiveness (efficacy and safety) of levetiracetam (LEV) versus the 2 older antiepileptic drugs (AEDs), sodium valproate extended release (VPA-ER) and carbamazepine controlled release (CBZ-CR) in the treatment of subjects with newly diagnosed epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy (all types of seizures) was made during the past year
* Subjects must have had at least two unprovoked seizures in the past 2 years with at least one during the last 6 months
* Female subjects without childbearing potential are eligible. Female subjects with childbearing potential are eligible if they use a medically accepted contraceptive method

Exclusion Criteria:

* Subjects previously allocated to a trial treatment (CBZ, VPA and LEV) used in this trial
* Participation in another clinical trial with an investigational drug or device within 12 weeks of the selection visit (V1), or at any time during this trial
* Pregnant or lactating women
* Presence of known pseudoseizures within the last year
* Uncountable seizures (clusters) or history of convulsive status epilepticus
* Any disorder or condition that may interfere with the absorption, distribution, metabolisation or excretion of drugs
* History of suicide attempt, current suicidal ideation, or other serious psychiatric disorders requiring or having required hospitalization or medication within the previous five years
* Presence of progressive cerebral disease, any other progressively degenerative neurological disease, or any cerebral tumors
* Presence of a terminal illness or any medical condition that might interfere with the subject's trial participation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1701 (Actual)
Dates: Start 2005-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Time to withdrawal from study medication (starting at V1) as a measure of combined efficacy and safety | Visit 1 to End of Study (approximately 52 weeks)

SECONDARY OUTCOMES:
The time to withdrawal comparing Levetiracetam versus the older Antiepileptic Drugs based on the subset of subjects whose best recommended treatment was Carbamazepine Controlled Release or Sodium Valproate Extended Release | Visit 1 to End of Study (approximately 52 weeks)
The retention rate after 6 months comparing Levetiracetam versus the older Antiepileptic Drugs | Visit 1 to Visit 4 (approximately 26 weeks)
The retention rate after 12 months comparing Levetiracetam versus the older Antiepileptic Drugs | Visit 1 to Visit 5 (approximately 52 weeks)
The retention rate after 6 months comparing Levetiracetam versus older Antiepileptic Drugs based on the subset of subjects whose best recommended treatment was Carbamazepine Controlled Release or Sodium Valproate Extended Release | Visit 1 to Visit 4 (approximately 26 weeks)
The retention rate after 12 months comparing Levetiracetam versus older Antiepileptic Drugs based on the subset of subjects whose best recommended treatment was Carbamazepine Controlled Release or Sodium Valproate Extended Release | Visit 1 to Visit 5 (approximately 52 weeks)
Seizure freedom at 6 months comparing Levetiracetam versus older Antiepileptic Drugs | Visit 1 to Visit 4 (approximately 26 weeks)
Seizure freedom at 12 months comparing Levetiracetam versus older Antiepileptic Drugs | Visit 1 to Visit 5 (approximately 52 weeks)
Seizure freedom at 6 months comparing Levetiracetam versus older Antiepileptic Drugs based on based on the subset of subjects whose best recommended treatment was Carbamazepine Controlled Release or Sodium Valproate Extended Release | Visit 1 to Visit 4 (approximately 26 weeks)
Seizure freedom at 12 months comparing Levetiracetam versus older Antiepileptic Drugs based on based on the subset of subjects whose best recommended treatment was Carbamazepine Controlled Release or Sodium Valproate Extended Release | Visit 1 to Visit 5 (approximately 52 weeks)
Time to first seizure comparing Levetiracetam versus older Antiepileptic Drugs | Visit 1 to End of Study (approximately 52 weeks)
Time to first seizure comparing Levetiracetam versus older Antiepileptic Drugs based on the subset of subjects whose best recommended treatment was Carbamazepine Controlled Release or Sodium Valproate Extended Release | Visit 1 to End of Study (approximately 52 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (229):
- Australia (12):
  - Adelaide
  - Bedford Park
  - Brisbane
  - Cairns
  - Camperdown
  - Chatswood
  - Clayton
  - Maroochydore
  - Parkville
  - Perth
  - Randwick
  - West Heidelberg
- Austria (6):
  - Graz
  - Innsbrick
  - Klagenfurt
  - Linz
  - Steyr
  - Vienna
- Belgium (10):
  - Bruges
  - Dendermonde
  - Edegem
  - Ghent
  - Haine-Saint-Paul
  - Jette
  - Kortrijk
  - Leuven
  - Ostend
  - Ottignies
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- Czechia (3):
  - Litomyšl
  - Ostrava-Poruba
  - Zlín
- Denmark (4):
  - Aalborg
  - Copenhagen
  - Holbæk
  - Holstebro
- Finland (3):
  - Hus (Helsinki)
  - Kuopio
  - Tampere
- France (25):
  - Blaye
  - Bordeaux
  - Brest
  - Carcassonne
  - Cherbourg
  - Colmar
  - Creil
  - Dijon
  - Freyming-Merlebach
  - Grenoble
  - La Seyne-sur-Mer
  - Lille
  - Lyon
  - Marseille
  - Mulhouse
  - Nancy
  - Nîmes
  - Paris
  - Rennes
  - Roanne
  - Saint-Brieuc
  - Saint-Quentin
  - Toulouse
  - Valenciennes
  - Vesoul
- Germany (37):
  - Altenburg
  - Arnsdorf
  - Aschaffenburg
  - Bamberg
  - Berlin
  - Bernau
  - Bernburg
  - Bielefeld
  - Bonn
  - Butzbach
  - Celle
  - Dillingen
  - Dresden
  - Düsseldorf
  - Erbach im Odenwald
  - Essen
  - Giessen
  - Göttingen
  - Halle
  - Hamburg
  - Hohenschönhausen
  - Jena
  - Königsbrück
  - Leipzig
  - Lengerich
  - Liegau-Augustusbad
  - Mittweida
  - Münster
  - Neukirchen-Vluyn
  - Neumünster
  - Oldenburg
  - Potsdam
  - Quickborn
  - Regenburg
  - Schalmstadt-Treysa
  - Siegen
  - Wermsdorf
- Greece (6):
  - Aklion
  - Alexandroupoli
  - Athens
  - Pátrai
  - Thessaloniki
  - Thessalonikis
- Hungary (3):
  - Budapest
  - Debrecen
  - Pécs
- Dublin, Ireland
- Italy (33):
  - Ancona
  - Asti
  - Bari
  - Busto Arsizio
  - Casarano
  - Catania
  - Cremona
  - Eboli
  - Faenza
  - Ferrara
  - Florence
  - Foggia
  - Forlì
  - Garbagnate
  - Grosseto
  - Milan
  - Napoli
  - Padua
  - Perugia
  - Pescara
  - Pisa
  - Potenza
  - Prato
  - Ragusa
  - Reggio Emilia
  - Roma
  - Siena
  - Taranto
  - Torino
  - Udine
  - Verona
  - Vimercate
  - Vittoria
- Netherlands (6):
  - Eindhoven
  - Heerenvegen
  - Leeuwarden
  - Maastricht
  - Nijmegen
  - Tilburg
- Norway (10):
  - Drammen
  - Fredrikstad
  - Lillehammer
  - Molde
  - Nordbyhagen
  - Sandvika
  - Stavanger
  - Tromsø
  - Trondheim
  - Tønsberg
- Poland (11):
  - Bydgoszcz
  - Częstochowa
  - Gdansk
  - Kielce
  - Krakow
  - Lodz
  - Lublin
  - Olsztyn
  - Poznan
  - Warsaw
  - Zgierz
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Craiova
- Russia (3):
  - Krasnoyasrk
  - Moscow
  - Saint Petersburg
- Slovakia (5):
  - Bratislava
  - Dolný Kubín
  - Dubnica nad Váhom
  - Martin
  - Žilina
- Spain (15):
  - Badalona
  - Barakaldo Vizcaya
  - Barcelona
  - Castellon
  - Elda
  - Girona
  - Leganes (Madrid)
  - Madrid
  - Móstoles
  - Murcia
  - Santa Cruz de Tenerife
  - Seville
  - Terrassa
  - Valencia
  - Vigo
- Sweden (5):
  - Karlstad
  - Linköping
  - Motala
  - Stockholm
  - Varberg
- Switzerland (6):
  - Bern
  - Biel
  - Geneva
  - Lausanne
  - Sankt Gallen
  - Zurich
- Turkey (Türkiye) (5):
  - Adana
  - Ankara
  - Bursa
  - Istanbul
  - Izmir
- United Kingdom (14):
  - Ashford
  - Bangor
  - Bristol
  - Cardiff
  - Dundee
  - Leeds
  - Liverpool
  - London
  - Plymouth
  - Southampton
  - Stoke-on-Trent
  - Sunderland
  - Swindon
  - Truro

REFERENCES:
- [Derived] Pohlmann-Eden B, Marson AG, Noack-Rink M, Ramirez F, Tofighy A, Werhahn KJ, Wild I, Trinka E. Comparative effectiveness of levetiracetam, valproate and carbamazepine among elderly patients with newly diagnosed epilepsy: subgroup analysis of the randomized, unblinded KOMET study. BMC Neurol. 2016 Aug 23;16(1):149. doi: 10.1186/s12883-016-0663-7. PMID 27552848
- [Derived] Trinka E, Marson AG, Van Paesschen W, Kalviainen R, Marovac J, Duncan B, Buyle S, Hallstrom Y, Hon P, Muscas GC, Newton M, Meencke HJ, Smith PE, Pohlmann-Eden B; KOMET Study Group. KOMET: an unblinded, randomised, two parallel-group, stratified trial comparing the effectiveness of levetiracetam with controlled-release carbamazepine and extended-release sodium valproate as monotherapy in patients with newly diagnosed epilepsy. J Neurol Neurosurg Psychiatry. 2013 Oct;84(10):1138-47. doi: 10.1136/jnnp-2011-300376. Epub 2012 Aug 29. PMID 22933814